CLINICAL TRIAL: NCT05533398
Title: Effect of Stress Ball Use on Anxiety in Haemodialysis Patients: A Single-blind Randomized Controlled Crossover Study
Brief Title: Stress Ball Use on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/014
Record Dates: First submitted 2022-09-03; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Stress; Anxiety; Hemodialysis Complication
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball use (Experimental): They were asked to use the ball for at least 10 minutes during the dialysis treatment and when they felt stressed or unwell at home/work.
  Interventions: Other: Stress ball use
- Control group (No Intervention): During the control condition, patients received standard care and did not use stress ball.

INTERVENTIONS:
Other: Stress ball use — They were asked to use the ball for at least 10 minutes during the dialysis treatment and when they felt stressed or unwell at home/work. Patients with arteriovenous fistula or arteriovenous graft were instructed to use the stress ball with the other hand, where there was no vascular access.
  Arms: Stress ball use

SUMMARY:
Stress management in dialysis patients plays a key role in reducing these negativities and in maintaining both physical and mental well-being. In dialysis patients, on the other hand, the effectiveness of stress ball use on comfort and stress was evaluated, and no study was found that evaluated its effect on anxiety.

DETAILED DESCRIPTION:
Stress ball is one of the non-pharmacological methods used to distract individuals when they consciously focus on a stimulus. With the squeezing of the ball, the nerves in the hands are stimulated and stimuli are sent to the limbic region of the brain, and these stimuli provide an acupressure effect. At the same time, it is the easiest and cheapest method that allows the mind to get away from stress and maintain the mental well-being of the person.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* On maintenance hemodialysis three times per week for four hours per session
* Able to communicate in Turkish
* Willing to participate to the study

Exclusion Criteria:

* Having any health problems related to the hand/arm to use the stress ball
* Patients who did not want to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Depression Level at 12 Dialysis Session | Up to 2 months
  It will be assessed two times with Hospital Anxiety and Depression Scale (HADS). Seven of the 14 questions measure anxiety and seven measure depression. Responses are scored in a four-point Likert format between 0-3. The lowest score that patients can get from both subscales is 0, and the highest score is 21. The cut-off points of the Turkish version of HADS were determined as 10 for the anxiety subscale and 7 for the depression subscale.
Change From Baseline Anxiety Level at 12 Dialysis Session | Up to 2 months
  It will be assessed two times with Hospital Anxiety and Depression Scale (HADS). Seven of the 14 questions measure anxiety and seven measure depression. Responses are scored in a four-point Likert format between 0-3. The lowest score that patients can get from both subscales is 0, and the highest score is 21. The cut-off points of the Turkish version of HADS were determined as 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687
- [Result] Ozen N, Cinar FI, Askin D, Mut D, Turker T. Nonadherence in Hemodialysis Patients and Related Factors: A Multicenter Study. J Nurs Res. 2019 Aug;27(4):e36. doi: 10.1097/jnr.0000000000000309. PMID 30720548
- [Result] Cantekin I, Tan M. The influence of music therapy on perceived stressors and anxiety levels of hemodialysis patients. Ren Fail. 2013;35(1):105-9. doi: 10.3109/0886022X.2012.736294. Epub 2012 Nov 15. PMID 23151089